CLINICAL TRIAL: NCT02671799
Title: Evaluation of the Minimally Invasive VenTouch™ System in the Treatment of Functional Mitral Valve Regurgitation (FMR): First-In-Man Continuation Study
Brief Title: Evaluation of the Minimally Invasive VenTouch™ System in the Treatment of Functional Mitral Valve Regurgitation (FMR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mardil Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VenTouch CT004
Record Dates: First submitted 2016-01-20; First posted 2016-02-02 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-02

CONDITIONS: Functional Mitral Regurgitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VenTouch System Implant (Experimental): The VenTouch System is indicated for patients who have moderately severe or severe functional mitral regurgitation (grade 3 or 4 MR).
  Interventions: Device: VenTouch System Implant

INTERVENTIONS:
Device: VenTouch System Implant — The VenTouch System is intended for use in the treatment of functional MR (FMR) in adults who are symptomatic despite optimal medical management. It is intended for subjects with FMR with essentially normal leaflet anatomy and motion, with mitral valve regurgitation attributable mainly to annular dilatation with or without papillary muscle displacement. It is not intended to treat structural defects/degeneration of the mitral valve. The VenTouch System is used to reshape the base of the heart to bring the mitral valve leaflets into better coaptation. By doing so, it brings the mitral valve leaflets closer, allowing proper closure of the valve, and reducing or eliminating MR. There is provision of support to the ventricular myocardium below the annulus as well as the annulus, so the VenTouch System may allow long-term ventricular remodeling with positive impact on the functionality of the mitral valve.

SUMMARY:
This is a prospective, multi-center, single-arm study to evaluate the VenTouch System for treatment of moderate to moderate-severe functional mitral valve regurgitation [FMR].

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, single-arm First-In-Man Continuation study to evaluate safety and efficacy of the VenTouch System for treatment of subjects with functional MR enrolling up to 15 subjects who have been diagnosed with Grade 3-4 functional mitral valve regurgitation. The duration of the study follow-up is 36 months from the time of therapy adjustment. Data from this trial may be utilized in support of a CE study in Europe and/or a pilot IDE study in the U.S. Follow-up testing will be performed at 1 month, 3 months, 6 months, and 12, 24, and 36 months post-therapy adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. Symptomatic FMR of grade moderately severe to severe (3 to 4) with structurally normal leaflets (preferably with echocardiographic evidence of EROA> 0.20 cm2)
3. NYHA Class II to IV
4. Left Ventricular Ejection Fraction (LVEF) 20%-50%
5. Treatment with optimal guideline-directed medical therapy for heart failure for at least 30 days. Subjects must be receiving a beta blocker for 3 months and an ACE-I or ARB for one month unless, in the investigator's opinion, the subject is intolerant to beta blockers, ACE-I or ARB. Beta blockers and ACE-I (or ARB) doses should be stable for one month prior to study entry. Stable is defined as no more than a 100% increase or a 50% decrease in dose.
6. Subjects with a Class I indication for CRT implant according to current guidelines should have CRT implant prior to entry into the study. Subjects who have existing CRT implants may be included in the study if the implant has been in place for at least 90 days.
7. Left Ventricular End Diastolic Diameter (LVEDD) of 55 to 80 mm as determined by transthoracic echocardiography.
8. Subject is willing and available to return for study follow-up
9. Subject or legal representative understands and provides signed informed consent for participation in study
10. Acceptance of subject for trial enrollment after review of all subject baseline data by Study Selection Committee

Exclusion Criteria:

1. Life expectancy of less than 12 months due to conditions other than cardiac status
2. Identified need for any cardiovascular surgery
3. Untreated clinically significant coronary artery disease
4. Any procedure, condition or cardiac anatomy that may impact or compromise the pericardial space (e.g. prior mitral valve surgery, CABG, epicardial pacing leads, pericarditis, or other procedure involving pericardial access)
5. Percutaneous coronary intervention, acute coronary syndrome (e.g. STEMI or non-STEMI myocardial infarction, unstable angina) or clinically significant cardiac events (e.g hypotension, syncope, arrhythmias, embolism, heart failure exacerbation or any hospitalization) within 30 days of enrollment
6. Thoracic or cardiac surgery contraindication (e.g., acute respiratory distress, endocarditis, myocarditis, pericarditis)
7. Significant structural abnormality of the mitral valve (e.g. flail leaflets, ruptured or elongated chordae, prolapsed valve, perforated valve leaflets, significant calcification in the annulus, or calcification in the leaflets that restricts motion)
8. Severe symptomatic carotid stenosis
9. Severe or sustained pulmonary hypertension, defined by resting pulmonary artery systolic (PAS) pressure greater than or equal to 70 mm Hg
10. Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction
11. Hypotension (systolic pressure <90mm Hg)
12. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, or any other structural heart disease causing heart failure other than dilated cardiomyopathy
13. UNOS status 1 heart transplantation
14. Creatinine > 2.5 mg/dL (221 µmol/L) and/or renal failure requiring dialysis
15. Active systemic infection or bleeding
16. Autoimmune disorders and/or the use of immune suppression therapy
17. Females who are pregnant (as documented by HCG beta pregnancy test in females of child-bearing age) or lactating
18. Currently enrolled in another investigational drug or device study

Intra-Operative Exclusion Criteria:

1. Subjects with heart size outside of the offered VenTouch System size range
2. Significant structural abnormality of the mitral valve (e.g. flail leaflets, ruptured or elongated chordae, prolapsed valve, perforated valve leaflets, significant calcification in the annulus, or calcification in the leaflets that restricts motion)
3. Signs/indications of ischemia
4. Intra-operative coronary angiography demonstrates that there is compression of the coronary arteries or reduction in coronary blood flow due to the VenTouch implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate mean reduction in MR, and freedom from grade 3 and 4 MR at 6 months post-therapy adjustment, as measured by an echocardiographic core lab | 6 months
Evaluate Serious Adverse Event (SAE) rates at 6 months post-therapy adjustment | 6 months

SECONDARY OUTCOMES:
Evaluate Serious Adverse Event (SAE) rates | Through 36 Months
Evaluate mean reduction in MR, and freedom from grade 3 and 4 MR, as demonstrated by quantitative measures, as measured by an echocardiographic core lab | Through 36 Months
Quantitative assessment of reverse remodeling based on change in LVEDD, LVEF, as measured by an echocardiographic core lab | Through 36 Months
Improvement in patient symptoms as assessed by the NYHA functional class | Through 36 Months
Improvement in Six-Minute Walk | Through 36 Months
Improvement in Minnesota Living with Heart Failure Questionnaire | Through 36 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Na Homolce Hospital, Prague, Czechia
- Bordeaux Heart University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Sponsor Website — http://www.mardil.com/